CLINICAL TRIAL: NCT07359937
Title: Design of a Multicomponent Intervention to Reduce the Risk of Exposure to High Concentrations of Fluoride in Children in Huila, Colombia
Brief Title: Design of a Multicomponent Intervention to Reduce the Risk of Exposure Fluorine
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Antonio Nariño (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UAN-Fluorine
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Fluorosis, Dental; Fluorosis
Keywords: Fluorine; Fluorides; Enamel fluorosis; Primary prevention; Health education
MeSH Terms: conditions — Fluorosis, Dental; Fluoride Poisoning; Health Education

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Side (Experimental): multicomponent intervention
  Interventions: Behavioral: multicomponent intervention
- Control side (Active Comparator): Conventional intervention
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: multicomponent intervention — 1. Installation of physical barriers: a reverse osmosis water filter. 2. Educational sessions for parents: three thematic modules. 3. Educational sessions for children: one thematic modules. 4. Outreach activities: To ensure the sustainability of the intervention. 5. Maintenance phase: The population will have free access to educational resources through the "Camaleón Sonriente cuida tus dientes" (Smiling Chameleon Takes Care of Your Teeth)
  Arms: Experimental Side
Behavioral: Conventional intervention — The intervention will include training on the cariogenic diet, flossing, and hand washing.
  Arms: Control side

SUMMARY:
Introduction Systemic exposure to fluoride is a significant challenge for global public health; this is because although fluoride prevents dental caries, prolonged exposure to high concentrations can cause adverse effects on various organs and systems, especially the teeth. Despite the existence of preventive strategies to reduce this exposure, evidence on the effectiveness of multicomponent interventions is limited. This protocol describes the design of a randomized controlled trial to evaluate the effects of a multicomponent intervention on parents and children to reduce the risk of exposure to high concentrations of fluoride in children. Methods This is a randomized controlled trial, and kindergartens in the municipalities of the Department of Huila, Colombia, will be recruited. The intervention group will receive a comprehensive five-component program: installation of water filters to reduce fluoride consumption; educational sessions for parents and children to raise awareness and promote healthy practices; outreach activities to strengthen collective knowledge; and a maintenance phase to ensure the program's sustainability. In contrast, the control group will participate in a conventional educational strategy focused on the parent-child dyad. Measurements will be taken at four points in time: pre-intervention for baseline and post-intervention at 3, 6, and 12 months. The evaluation of results includes the concentration of fluoride in children's urine, fluoride levels in water (to validate the effectiveness of filtration), and changes in parents' knowledge, attitudes, and practices. Discussion The trial will evaluate the effectiveness of a multicomponent intervention aimed at parents and children to reduce the risk of fluoride exposure. Through integrative methodological approaches and objective measurements, it will demonstrate significant improvements in reducing fluoride exposure in children and in parents' knowledge, attitudes, and practices. It will contribute to child health programs, strengthen preventive oral health strategies with an impact on public policy, community health, and new lines of research on fluoride.

ELIGIBILITY:
Inclusion Criteria:

* Kindergartens located in municipalities with exposure to fluoride concentrations in water.
* Have a school feeding program.
* The child must be enrolled.
* They must be registered in the school feeding program.
* The primary caregiver must be able to read.
* The caregiver must agree to participate voluntarily and sign the informed consent form.
* The caregiver must commit to attending all components of the intervention (education and collection of the child's urine sample).

Exclusion Criteria:

* Parents or children with conditions or situations that may interfere with the assimilation of the components of the strategy.
* Children who wear diapers will be excluded from the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Urinary fluoride concentrations | Time Frame: Baseline, 3 , 6, and 12 months.
  Decrease in urinary fluoride concentrations in children

SECONDARY OUTCOMES:
Knowledge, attitudes, and practices (KAP) | Time Frame: Baseline, 3 , 6 and 12 months.
  To assess changes in parents' knowledge and attitudes, the Knowledge, Attitudes, and Practices (KAP) survey will be administered, after validation. The instrument was designed for this purpose, taking into account the components of the intervention. The knowledge section consists of 12 items and explores parents' understanding of natural and non-natural sources of fluoride and its effects on oral and systemic health. The attitudes section consists of 10 items and identifies perceptions, beliefs, motivations, and willingness to act in response to fluoride risk, water quality, willingness to change habits, and dental follow-ups. The practices section, with 9 items, addresses information on current behaviors related to consulting fluoride content, modifying water sources, dental care, and supervision in the use of dental products. Each section of the instrument includes ordinal scale variables and provides an overall score that allows each section to be classified as good, fair, or poor.
Fluoride concentrations in water | Time Frame: baseline, 3, 6, and 12 months
  Reduction in fluoride concentrations in water.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de desarrollo infantil - Sonrisitas de oro, Palermo, Colombia